CLINICAL TRIAL: NCT01092299
Title: A Phase I Study to Investigate the Relative Bioavailability of Modified-release Formulations of AZD1446 Compared to an Immediate-release Capsule Under Fed and Fasting Conditions Following Single and Repeated Dose Administration to Young and Elderly Healthy Volunteers
Brief Title: A Bioavailability Study Comparing Modified-release Capsules and Immediate Release Capsules in Fed and Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D1950C00008; 2009-017702-36 (EudraCT Number)
Record Dates: First submitted 2010-03-10; First posted 2010-03-24 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Phase I; Relative bioavailability; Pharmacokinetic study; AZD1446; healthy volunteers
MeSH Terms: interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (2 arms) (Experimental): Period 1: randomized to either fasting IR or ER1. Period 2: Cross-over to either IR or ER1. Period 3: ER1 in fed conditions.
  Interventions: Drug: AZD1446
- Cohort 2 (2 arms) (Experimental): Period 1: randomized to either fasting IR or ER2. Period 2: Cross-over to either IR or ER2. Period 3: ER2 in fed conditions.
  Interventions: Drug: AZD1446
- Cohort 3( 2 arms) (Experimental): Period 1: randomized to either fasting IR or ER3. Period 2: Cross-over to either IR or ER3. Period 3: ER3 in fed conditions.
  Interventions: Drug: AZD1446
- Cohort 4 (2 arms) (Experimental): Period 1: randomized to either fasting IR or MR4. Period 2: Cross-over to either IR or MR4. Period 3: MR4 in fed conditions.
  Interventions: Drug: AZD1446
- Part 2: Extended/Modified release (Experimental): Extended/Modified release capsule to be determined
  Interventions: Drug: AZD1446
- Part 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1446 — ER Fast, 90mg, p.o. capsule
  Arms: Cohort 1 (2 arms)
Drug: AZD1446 — ER Moderate, 90mg, p.o. capsule
  Arms: Cohort 2 (2 arms)
Drug: AZD1446 — ER Slow, 90mg, p.o. capsule
  Arms: Cohort 3( 2 arms)
Drug: AZD1446 — MR
  Arms: Cohort 4 (2 arms); Part 2: Extended/Modified release
Drug: AZD1446 — IR, 90 mg p.o. capsule
  Arms: Cohort 4 (2 arms); Part 2: Extended/Modified release
Drug: Placebo — IR
  Arms: Part 2: Placebo
Drug: Placebo — ER/MR
  Arms: Part 2: Placebo

SUMMARY:
Part 1: The purpose of this study is to determine the pharmacokinetic profile of 4 different Extended/modified-release formulations and one immediate release formulation of AZD1446. In addition the food effect on AZD1446 pharmacokinetics will be investigated.

Part 2: To asses the safety and tolerability of the selected formulation(s) from part 1 in elderly healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 19 and 30 kg/m2
* Clinically normal findings on physical examination

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* History or present symptoms or signs of severe allergy/hypersensitivity reactions including severe food allergy, as judged by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Part 1: Single Dose Administration :• Cmax, tmax, t½λz, AUC0-t, AUC, AUC0-τ (Part 2 only), Frel (Part 1 only), CL/F, Vz/F | Part 1 - 11 days
Part 2 Multiple Dose Administration: - Cmax, tmax, t½λz, AUC0-t, AUC, AUC0-τ (Part 2 only), Frel (Part 1 only), CL/F, Vz/F Day 9 of Part 2 following multiple dosing in addition to the above • Cmin, tmin, Cavg, fluctuation ratio, RCmax, RAUC(0-τ) | Part 2 - 10 days

SECONDARY OUTCOMES:
Part 1: Safety and tolerabilty :- Laboratory safety data, vital signs, electrocardiogram, Columbia-Suicide Severity Rating Scale, adverse events, Mini-international neuropsychiatric interview | throughout the approx 7 weeks of study duration
Part 1: Single Dose Administration :• Cmax, tmax, t½λz, AUC0-t, AUC, AUC0-τ (Part 2 only), Frel (Part 1 only), CL/F, Vz/F | Part 1 - 11 days
Part 2 Multiple Dose Administration :- Cmax, tmax, t½λz, AUC0-t, AUC, AUC0-τ (Part 2 only), Frel (Part 1 only), CL/F, Vz/F Day 9 of Part 2 following multiple dosing in addition to the above • Cmin, tmin, Cavg, fluctuation ratio, RCmax, RAUC(0-τ | Part 2 - 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Lena Bolin, Study Director — AstraZeneca R&D; Aslak Rautio, Principal Investigator — Quintiles Hermelinen AB; Wolfgang Kühn, Principal Investigator — Quintiles AB, Phase I Services
Locations (2):
- Sweden (2):
  - Research Site, Luleå
  - Research Site, Uppsala